CLINICAL TRIAL: NCT05948644
Title: Phase Ib Clinical Study on the Safety, Tolerability, and Pharmacokinetics of TPN171H Tablets in the Treatment of Pulmonary Arterial Hypertension (PAH) Patients
Brief Title: The Safety, Tolerability, and Pharmacokinetics of TPN171H Tablets in Patients With Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Collaborators: Shanghai Institute of Materia Medica, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPN171H-04
Record Dates: First submitted 2023-06-21; First posted 2023-07-17 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TPN171H (Experimental): TPN171H is received 2.5mg QD for 2 consecutive weeks, then 5 mg QD for 14 consecutive weeks. If the dose is well-tolerated,TPN171H is up-titrated to 10mg QD , which will last for up to 2 years.
  Interventions: Drug: TPN171H

INTERVENTIONS:
Drug: TPN171H — TPN171H 2.5mg TPN171H 5mg TPN171H 10mg

SUMMARY:
Exploring the safety, tolerability, and pharmacokinetic (PK) characteristics of oral TPN171H tablets in patients with Pulmonary Arterial Hypertension under continuous multiple administration conditions, providing a basis for determining the administration plan and recommended dosage in phase II clinical study.

DETAILED DESCRIPTION:
This study was divided into screening period, treatment period and medication follow-up period, and the treatment period included 3 cycles.

First cycle: subjects receiving the test drug 2.5mg QD for 2 consecutive weeks, PK blood collection on Day 1 and Day 7, and the subjects discharged and returned to the hospital on Day 14 for medication monitoring blood collection, safety examination and efficacy assessment.

Second cycle: up to 14 weeks; the second cycle is divided into monitoring and observation cycles; subjects who complete the first cycle and examinations enter the second cycle, with a 14 day monitoring period and 12 week observation period, with the second cycle dose of 5 mg QD, subjects received PK sampling on Day 7.

Third cycle:The third cycle lasts for 8 days, subjects receive 10mg QD for 8 days; subjects received PK sampling on Day 7; subjects who completed an 8-day safety observation period on Day 8 without abnormal safety tests may be discharged. After discharge into the medication follow-up period.

Medication follow-up period: up to 2 years; subjects entering the follow-up period will continue to take the dose of the last treatment period, return to hospital once every 12 weeks for safety examination and efficacy assessment until the subject intolerance or withdrawal from the study or expiration of 2 years (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are able to signed the informed consent form ,understand and follow study plans and instructions;
2. Patients aged 18 to 75;
3. Patients with symptomatic PAH (Group1) with right heart catheterization results within the past 36 months (first category), a pulmonary vascular resistance (PVR) > 3 Wood, a mean pulmonary artery pressure (mPVP) ≥25 mmHg and a pulmonary artery wedge pressure (PAWP) ≤ 15 mmHg ;
4. Patients have a current diagnosis of being in WHO functional class II or III;
5. Targeted therapeutic drugs were not added, discontinued, or dosed within 4 weeks prior to baseline; 6.6-MWD between 100m &450m;

7.Patients who are willing to take proper contraceptive during the study and within 3 months after the study completed.

Exclusion Criteria:

1. All types of PH except subtypes of Group1 specified in the inclusion criteria;
2. Patients who concomitant severe obstructive pulmonary disease(FEV1/FVC<0.5) ;
3. Total lung volume<60% predicted;
4. Systolic blood pressure below 90/60mmHg at screening;
5. Left ventricular ejection fraction less than 45%, left ventricular short axis shortening rate less than 0.2;
6. Lower limb diseases that affect the completion of 6-MWD testing;
7. Subjects who received PDE5 inhibitors (such as sildenafil, tadalafil, vardenafil, and avanafil) within 4 weeks before baseline
8. CYP3A4 enzyme inducers (such as bosentan, aprepitant, barbiturates, carbamazepine, rifampicin, pioglitazone) or inhibitors (such as cimetidine, ciprofloxacin, boceprevir-d9，telaprevir, clarithromycin, nefazodone, and ritonavir) were taken within 2 months before the start of the trial, Regular or intermittent administration of nitrates (such as nitroglycerin, isosorbide nitrate,pentaerithrityl tetranitrate ) or any form of nitric oxide donor (including nicorandil, L-arginine) and α- Receptor blocking (such as phenoxybenzamine, prazosin, terazosin,tamsulosin)
9. Subjects with a clear history of allergic diseases or who have previously stopped taking either aniracetam or tadalafil due to safety or tolerable reasons;
10. Previous or current drug dependence, clear history of neurological or mental disorders, such as epilepsy, dementia, psychological or other emotional issues, may invalidate informed consent or limit the subject's ability to comply with the protocol;
11. Acute or chronic organic diseases (excluding breathing difficulties) prevent subjects from completing the necessary testing items required in the study (especially the 6-minute walking distance test);
12. Have a history of ophthalmic diseases, such as color vision abnormalities, retinitis pigmentosa, and macular degeneration;
13. Malignant tumor patients;
14. Moderate or severe liver function injury and/or blood ALT and AST exceeding 1.5 times the upper limit of normal values, and blood creatinine exceeding 1.5 times the upper limit of normal values;
15. Pathogenic test for HIV positive; Positive test for hepatitis B or hepatitis C; Subjects suffering from acute infectious diseases;
16. Suffered from infectious diseases recently (within 1 month);
17. The subject has ischemic heart disease (defined as symptomatic, requiring anti angina treatment, or having experienced myocardial infarction within the past 3 years);
18. Those who have experienced cerebrovascular events (such as transient ischemic attacks or strokes) within the past 3 months;
19. Participated in any clinical trial within 3 months prior to taking the investigational drug;
20. Pregnant or lactating women;
21. The researchers believe that subjects who are not suitable to participate in this experiment due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | through study completion, an average of 2 years
Q-T interval | through study completion, an average of 2 years
Tmax | From time zero up to 24 hours post-dose following oral administration of TPN171H
Cmax | From time zero up to 24 hours post-dose following oral administration of TPN171H
AUC0~t | From time zero up to 24 hours post-dose following oral administration of TPN171H
AUC0-∞ | From time zero up to 24 hours post-dose following oral administration of TPN171H
Terminal half-life (t 1/2) | From time zero up to 24 hours post-dose following oral administration of TPN171H
Apparent distribution volume (Vd/F) | From time zero up to 24 hours post-dose following oral administration of TPN171H
Clearance rate (CL/F) | From time zero up to 24 hours post-dose following oral administration of TPN171H
Mean Residence Time(MRT) | From time zero up to 24 hours post-dose following oral administration of TPN171H

SECONDARY OUTCOMES:
6- Minute Walk Distance（6-MWD） | through study completion, an average of 2 years
  Cardiopulmonary function indicators reflecting the patient's physiological state
NT-proBNP | through study completion, an average of 2 years
  Heart failure evaluation indicators to evaluate the severity of heart failure;
The World Health Organization (WHO) functional class | through study completion, an average of 2 years
  Evaluate the severity of Pulmonary Arterial Hypertension symptoms at each time point before and after taking TPN171H
Borg dyspnea index | through study completion, an average of 2 years
  to evaluate the degree of difficulty breathing in subjects after a 6-minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Fu Zhu, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Fu Zhu, Shanghai, China

IPD SHARING:
Plan to Share IPD: No